CLINICAL TRIAL: NCT04124302
Title: The Impact of Two Different Insulin Dose Calculation on Postprandial Glycemia After Mixed Meal in Children With Type 1 Diabetes Mellitus- Randomized Study.
Brief Title: The Impact of Two Different Insulin Dose Calculation on Postprandial Glycemia After Mixed Meal.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Mixed Meal Bolus
Record Dates: First submitted 2019-08-23; First posted 2019-10-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes type 1; insulin bolus; prandial insulin requirement; postprandial glycemia; insulin pump therapy; mixed meal
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine; Insulin Aspart; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPF (Active Comparator): Total meal bolus will consist of insulin for carbohydrates (IC) and insulin for proteins and fats (IPF) based on individual insulin-to-carbohydrate ratio (ICR). Dual bolus will be given 15 minutes before the mixed meal (toast with cheese).
  Interventions: Drug: Insulin Glulisine; Drug: Insulin Aspart; Drug: Insulin Lispro
- 30%IC (Experimental): Total meal bolus will consist of insulin for carbohydrates (IC) calculated based on individual insulin-to-carbohydrate ratio (ICR) and insulin for proteins and fats (IPF) estimated as 30% of IC. Dual bolus will be given 15 minutes before the mixed meal (toast with cheese).
  Interventions: Drug: Insulin Glulisine; Drug: Insulin Aspart; Drug: Insulin Lispro

INTERVENTIONS:
Drug: Insulin Glulisine — A kind of bolus insulin will be insulin glulisine if participant used insulin glulisine before entering the trial.
  Other Names: Apidra
Drug: Insulin Aspart — A kind of bolus insulin will be insulin aspart if participant used insulin aspart before entering the trial.
  Other Names: NovoRapid
Drug: Insulin Lispro — A kind of bolus insulin will be insulin lispro if participant used insulin lispro before entering the trial.
  Other Names: Humalog, Liprolog

SUMMARY:
The aim of the study is to compare the impact of two different insulin dose calculation on postprandial glycemia after mixed meal in children with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* duration of type 1 diabetes longer than 12 months
* insulin pump therapy longer than 3 months
* treated by the same type of insulin longer than 3 months
* written informed consent by patients and parents

Exclusion Criteria:

* celiac disease
* diabetes related complications (e.g. nephropathy)
* any disease judged by the investigator to affect the trial
* withdrawal of consent to participate in the study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemia | 30 minutes after meal
  Postprandial blood glucose excursion measured by self monitoring of blood glucose (SMBG).
Postprandial glycemia | 60 minutes after meal
  Postprandial blood glucose excursion measured by self monitoring of blood glucose (SMBG).
Postprandial glycemia | 90 minutes after meal
  Postprandial blood glucose excursion measured by self monitoring of blood glucose (SMBG).
Postprandial glycemia | 120 minutes after meal
  Postprandial blood glucose excursion measured by self monitoring of blood glucose (SMBG).
Postprandial glycemia | 150 minutes after meal
  Postprandial blood glucose excursion measured by self monitoring of blood glucose (SMBG).
Postprandial glycemia | 180 minutes after meal
  Postprandial blood glucose excursion measured by self monitoring of blood glucose (SMBG).
Postprandial glycemia | 210 minutes after meal
  Postprandial blood glucose excursion measured by self monitoring of blood glucose (SMBG).
Postprandial glycemia | 240 minutes after meal
  Postprandial blood glucose excursion measured by self monitoring of blood glucose (SMBG).
Postprandial glycemia | 270 minutes after meal
  Postprandial blood glucose excursion measured by self monitoring of blood glucose (SMBG).
Postprandial glycemia | 300 minutes after meal
  Postprandial blood glucose excursion measured by self monitoring of blood glucose (SMBG).

SECONDARY OUTCOMES:
Glucose Area Under the Curve (AUC) | 5 hours study period
  Measurements based on Continuous Glucose Monitoring System (CGMS)
The Difference Between The Maximum and Baseline Glucose Level - mean amplitude of glycaemic excursion (MAGE) | 5 hours study period
  Measurements based on SMBG
Hypoglycemia Episodes | 5 hours study period
  Hypoglycemia defined as a plasma glucose concentration below 70mg/dl with or without symptoms
Time in target postprandial glycemia | 5 hours study period
  Time spent in the target range between 70 and 180 mg/dL based on CGMS

CONTACTS AND LOCATIONS:
Locations (1):
- Warsaw Medical University, Warsaw, Poland